CLINICAL TRIAL: NCT03812081
Title: A Comparative Study of the Baska Mask Vs Proseal Laryngeal Mask Regarding Airway Sealing Pressure According to Confirmation by Fiberoptic Position
Brief Title: A Comparative Study of the Baska Mask Vs Proseal Laryngeal Mask Regarding Airway Sealing Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N_50_2018
Record Dates: First submitted 2019-01-11; First posted 2019-01-22 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Baska Mask

STUDY DESIGN:
Intervention Model Description: Following approval from EL Kasr Al-Ainy teaching hospital ethical committee and an informed patient consent, the investigators enrolled 74adult patients ASA I and II, non-obese (BMI<30) ranging from18-45 yrs. of age, Patients underwent a variety of elective surgical procedures in the supine position with SAD placement for ≤ 2 hours duration. Patients randomly divided by computer designed lists and then concealed in closed envelopes into 2 equal groups:
  Group A (n= 37), in which Baska Mask Airway _ (size 3,4,5) will used for ventilation according of patient body weight.
  Group B (n= 37), in which Laryngeal Mask Airway- Proseal LMA_ (size 3,4,5) was used for ventilation according of patient body weight.
Who Masked: Participant, Care Provider
Masking Description: 72 Patients are randomly divided by computer designed lists and then concealed in closed envelopes into 2 equal groups: Group A (n= 37), in which Baska Mask Airway _ (size 3,4,5) will used for ventilation according of patient body weight.
  Group B (n= 37), in which Laryngeal Mask Airway- Proseal LMA_ (size 3,4,5) was used for ventilation according of patient body weight
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Baska Mask (Active Comparator): In which Baska Mask Airway (size 3,4,5) will used for ventilation according of patient body weight.Size selection is based on the manufacturer's recommendation of weight-based estimate plus clinical judgment. The Baska Mask is available in four sizes: size three (30 to 50 kg), size four (50 to 70 kg), size five (70 to 100 kg),The membranous cuff of the Baska Mask appears bulkier than the equivalent inflatable cuff on cuffed laryngeal masks. The mask can easily be decreased in size during insertion by compressing the proximal, firmer part of the mask below the airway tube, between the thumb and two fingers
  Interventions: Device: Group A : Baska Mask Airway
- Group B Proseal Mask (Active Comparator): In which Laryngeal Mask Airway- Proseal LMA (size 3,4,5) was used for ventilation according of patient body weight.Size selection is based on the manufacturer's recommendation of weight-based estimate plus clinical judgment.
  Interventions: Device: Group B: Proseal Laryngeal Mask Airway

INTERVENTIONS:
Device: Group A : Baska Mask Airway — Size selection is based on the manufacturer's recommendation of weight-based estimate plus clinical judgment. The Baska Mask is available in four sizes: size three (30 to 50 kg), size four (50 to 70 kg), size five (70 to 100 kg),The membranous cuff of the Baska Mask appears bulkier than the equivalent inflatable cuff on cuffed laryngeal masks. The mask can easily be decreased in size during insertion by compressing the proximal, firmer part of the mask below the airway tube, between the thumb and two fingers
  Arms: Group A Baska Mask
Device: Group B: Proseal Laryngeal Mask Airway — Proseal LMA (size 3,4,5) was used for ventilation according of patient body weight.Size selection is based on the manufacturer's recommendation of weight-based estimate plus clinical judgment.
  Arms: Group B Proseal Mask

SUMMARY:
Baska mask air way(BM) in comparative study with Proseal laryngeal mask airway (PLMA) regarding performance of Baska mask improves the safety and efficacy of airway management for in patients undergoing general anesthesia by mechanical ventilation confirmation of position by fiber optic view of glottis opening and success of gastric tube insertion , Airway sealing pressure, Leak fraction, insertion time and "overall insertion" success rates, and post-operative complications (airway trauma, hoarseness, sore throat and Dysphagia ).

DETAILED DESCRIPTION:
Maintenance of a patent airway is a major responsibility for the anesthesiologists, interruption of gas exchange, even for a few minutes, can result in catastrophic outcomes such as brain damage or death.

Supraglottic airway devices are devices that ventilate patients by delivering anaesthetic gases/oxygen above the level of the vocal cord. Since the development of the laryngeal mask airway, many other supraglottic devices have been introduced in the clinical practice of airway management, trying to offer a simple and effective alternative to endotracheal tube.

However, following experience with such simple cases, clinicians soon become comfortable with more complex cases, such as cases of longer duration, cases with sicker patient reported favorable outcomes in safety profile, risk, ease of insertion, recovery of patients and cost analyses. However, there is an under reporting of complications aris¬ing during ventilation with this device and the risk factors associated with such complications in adult patients. These include Hypoxia, laryngospasm, and difficulty with insertion, suboptimal ventilation, bronchospasm, aspiration, desaturation, hy¬potension and conversion to intubation with ETT. These can be significantly serious and life threatening

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult ASA I-II patients,
2. Both genders, aged 18-45 years,
3. Body weight between 50 and 90 kg who BMI > 30 kg/m2
4. Non-urgent surgery of planned duration up to 2 hrs

Exclusion Criteria:

1. Patient refusal
2. Patients having known tendency to nausea/vomiting or pharyngeal pathology
3. Morbid obese patients with body mass index >30 kg/m2
4. Patients known to have gastro-esophageal reflux disease (GERD), hiatus hernia or previous upper gastrointestinal tract surgery
5. History of difficult intubation, measured the common predictive indices for difficult intubation (BMI, thyromental distance,Mallampati grade, inter-incisor distance, dentition and neck movement ).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Airway sealing pressure in cmH2O | 15 Minutes
  The airway sealing pressure is the pressure at which leak starts; in cmH2O at 5 mints post placement, this leak pressure will calculate as the plateau airway pressure reach with fresh gas flow 6 l/min, and pressure adjustment valve set at 70 cmH2O, and observing of the rise of the ventilator's airway pressure.
  A ''puffing'' sound was heard near the patient's mouth (release of pressure) indicating the airway seal pressure

SECONDARY OUTCOMES:
Laryngeal view grades recorded by fiberoptic bronchoscopes. | 15 Minutes
  fiberoptic bronchoscopes can record Laryngeal view grades
Device Complications: | Through study completion
  Patients will be monitoring for the following complications: arterial oxygen desaturation, lip damage; blood staining on mask removal and laryngospasm, the incidence and severity of throat pain, dysphagia, Heart burn, Nausea and Vomiting at arrival and discharge from the recovery unit and on the first postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Press